CLINICAL TRIAL: NCT04418024
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of AG10 in Subjects with Symptomatic Transthyretin Amyloid Polyneuropathy (ATTRibute-PN Trial)
Brief Title: Efficacy and Safety of AG10 in Subjects with Transthyretin Amyloid Polyneurophathy
Acronym: ATTRibute-PN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: After a careful review of the currently available treatments worldwide for patients with ATTR-polyneuropathy, Eidos has made the decision to halt the current study design.
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG10-333; 2018-004670-10 (EudraCT Number)
Record Dates: First submitted 2020-05-22; First posted 2020-06-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-06

CONDITIONS: Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy
Keywords: TTR; ATTR-PN; Familial ATTR-PN; Amyloidosis; Amyloid; Transthyretin; Polyneuropathy; TTR-mediated amyloidosis; Amyloidosis, hereditary; Familial Amyloid Polyneuropathies; Amyloidosis, Hereditary, Transthyretin-Related
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis; Alzheimer Disease; Polyneuropathies; Amyloidosis, Familial; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AG10 800 mg (Experimental): TTR stabilizer administered orally twice daily (BID)
  Interventions: Drug: AG10
- Placebo (Placebo Comparator): Placebo administered orally twice daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AG10 — TTR stabilizer administered orally twice daily (BID)
  Other Names: Oral AG10
  Arms: AG10 800 mg
Drug: Placebo — Non-active control
  Other Names: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
See updated study design under NCT04882735. Phase 3 efficacy and safety of AG10 compared with placebo in subjects with symptomatic Transthyretin Amyloid Polyneuropathy (ATTR-PN)

DETAILED DESCRIPTION:
** See updated study design under ClinicalTrials.gov Identifier NCT04882735. **

Transthyretin amyloid polyneuropathy (ATTR-PN), also called "Familial Transthyretin-Mediated Amyloid Polyneuropathy (FAP)" is a hereditary condition caused by mutations in the TTR gene. It is estimated that around 10,000 people in the world are affected.

In ATTR-PN, amyloid builds up in the nerves that detect temperature, pain, and touch. Patients with ATTR-PN can experience a loss of sensation, tingling, numbness, or pain in the hands and feet (also called peripheral neuropathy).

In this study Eidos is researching the investigational drug AG10 800mg (2 tablets) administered orally twice a day. Through the study, Eidos wants to evaluate the efficacy and safety of AG10 in patients with ATTR-PN versus placebo.

This is an 18 month, placebo-controlled study. This means that, during the 18 month study, investigators conducting the research and study participants will not know whether the study participant is receiving AG10 or placebo.

The primary outcome of the study is the difference between AG10 and placebo groups in the Modified Neurologic Impairment Score +7 (mNIS+7) at 18 months of treatment versus baseline.

At the end of 18 months, participants may be eligible to receive investigational AG10, and there is no placebo. This is called an "open label extension." This part of the study may help us better understand the safety related to taking AG10 over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female ≥18 to ≤90 years of age;
* Have Stage I or II symptoms (polyneuropathy disability [PND] ≤IIIa) of ATTR-PN and an established diagnosis of ATTR-PN as defined by physical exam findings and/or neurophysiological test findings consistent with the diagnosis of ATTR-PN;
* Have an NIS of 5 to 130 (inclusive) during screening;
* Have a nerve conduction studies (NCS) score [sum of the sural sensory nerve action potential (SNAP), tibial compound muscle action potential (CMAP), ulnar SNAP, ulnar CMAP, and peroneal CMAP] of ≥2 points during screening. NCS is a component of mNIS+7;
* Have a mutation consistent with ATTR-PN either documented in medical history or confirmed by genotyping obtained at Screening prior to randomization. *No genetic testing is needed for subjects who are recipients of domino liver transplants;
* Have an anticipated survival of ≥2 years
* Have Karnofsky performance status ≥60 %;

Exclusion Criteria:

* Had a prior liver transplantation or is planning to undergo liver transplantation with a wild-type organ graft as treatment for symptomatic ATTR-PN during the study period.

Note: Recipients of a "domino" liver transplant from an ATTR-PN donor who have developed ATTR-PN mediated by their graft are allowed under this protocol, as long as re-transplantation to treat ATTR-PN is not planned during the study period and meets all other eligibility criteria;

* Has sensorimotor or autonomic neuropathy not related to ATTR-PN; for example, autoimmune disease or monoclonal gammopathy, malignancy, or alcohol abuse;
* Has Vitamin B-12 levels below the lower limit of normal (LLN);
* Has clinical evidence of untreated hyper/hypothyroidism;
* Has leptomeningeal TTR amyloidosis;
* Has Type 1 diabetes;
* Has had Type 2 diabetes for ≥5 years;
* Has active hepatitis B or C or known human immunodeficiency virus (HIV) infection;
* Has NYHA heart failure classification >Class II
* Had a malignancy within 2 years, except for basal or squamous cell carcinoma of
* Is currently undergoing treatment for ATTR-PN with patisiran, inotersen, or other gene silencing agents, marketed drug products lacking a label indication for ATTR- PN (e.g., diflunisal, doxycycline), natural products or derivatives used as unproven therapies for ATTR-PN (e.g., green tea extract, tauroursodeoxycholic acid [TUDCA]/ursodiol), within 14 days, or 90 days for patisiran and 180 days for inotersen prior to dosing. Prior to screening, tafamidis, if already prescribed to potential subjects as part of their established background therapy, is allowed at the labeled dosage and administration of 20 mg/day for the treatment of ATTR-PN with, i in the opinion of the Investigator, evidence of disease progression while on tafamidis treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Month 18 of treatment in Modified Neuropathy Impairment | 18 Months
  Evaluate the difference between the AG10 and placebo groups in Modified Neuropathy Impairment which is a composite scale that asses,in part, muscle weakness, sensory loss, and decreased muscle stretch reflexes. It is calculated on a scale of 0 to 304 with higher scores indicating a worsening of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mark McGovern, RN, CCRN, Study Director — Eidos Therapeutics, a BridgeBio company
Locations (1):
- Eidos Therapeutics, San Francisco, California, United States